CLINICAL TRIAL: NCT00459446
Title: Gadofosveset Imaging of Chronic Total Peripheral Artery Occlusion (CTO)
Brief Title: Imaging of Totally Blocked Arteries
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: NHLBI
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 070128; 07-H-0128
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-11-25

CONDITIONS: Atherosclerosis; Peripheral Artery Disease; Intermittent Claudication; Chronic Total Aterial Occlusion
Keywords: Magnetic Resonance Imaging; Gadolinium Contrast; Gadofosveset; Atherosclerosis; Chronic Total Arterial Occlusions; Cardiovascular Disease; Blocked Arteries; Peripheral Artery Disease; PAD; Intermittent Claudication; Chronic Total Arterial Occlusion
MeSH Terms: conditions — Atherosclerosis; Peripheral Arterial Disease; Intermittent Claudication; Cardiovascular Diseases | interventions — gadofosveset trisodium

INTERVENTIONS:
Drug: MS-325 Injection (Gadofosveset Trisodium)

SUMMARY:
This study will test how well a new contrast agent (dye) used in magnetic resonance imaging (MRI) can help visualize totally blocked arteries that normally supply blood to the neck, arms or legs. Currently used agents work well in visualizing normal or partly blocked arteries (arteries that have some blood flowing through them), but only poorly in totally blocked arteries. This study will see if a contrast agent called gadofosveset can better brighten images of completely blocked arteries. Gadofosveset is approved in Europe for use in MRI scans, but is still considered experimental in the United States.

People 18 years of age or older with known or suspected total blockage of an artery to the neck, arm or leg may be eligible for this study.

Participants undergo MRI scanning with gadofosveset contrast dye. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. For this procedure, the subject lies on a table that can slide in and out of the tubular scanner, wearing earplugs to muffle loud noises that occur during the scanning process. The procedure lasts about 1.5 to 2 hours, during which the subject may be asked to hold his or her breath several times for as long as 5 to 20 seconds. During the procedure, gadofosveset is injected and several kinds of MRI pictures are taken to understand better how the new agent works. Subjects may be asked to undergo a second scan using conventional MRI contrast dye

DETAILED DESCRIPTION:
Repairing totally occluded peripheral arteries remains challenging because they are not visualized using available imaging technologies. Contrast-enhanced magnetic resonance angiography (CE-MRA), X-ray computed tomography angiography (CTA), and invasive radiocontrast digital subtraction angiography (DSA) all rely on blood flow within arteries that are not totally occluded. Where the arterial lumen is totally occluded, contrast does not enter and the artery remains invisible. As a result, physicians have difficulty identifying a pathway or trajectory for catheter devices in order to improve blood flow using angioplasty.

Gadofosveset, an albumin-binding MRI contrast agent that is commercially available outside the United States, may accumulate in the walls of occluded arteries through a mechanism that is not known.

The goal of this protocol is to determine whether gadofosveset has value in planning catheter trajectories in totally occluded peripheral arteries. We propose to study the gadofosveset contrast enhancement patterns in occluded peripheral artery segments in up to 20 patients with known occluded iliac, femoral, and shoulder arteries being considered for catheter-based treatment.

This research may have value in planning and conducting minimally invasive treatments using conventional X-ray guidance and possibly in the future using investigational real-time MRI guidance.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects with known cardiovascular disease will be eligible for participation in this protocol. The subject is eligible under the following conditions:

* Subject's age is greater than 18 years of age.
* Known occlusion of iliac, femoral, or brachiocephalic arteries.

EXCLUSION CRITERIA:

Subjects with absolute contraindications to MRI scanning will be excluded. These contraindications include subjects with the following devices:

* Implanted cardiac pacemaker or defibrillator.
* Central nervous system aneurysm clips.
* Implanted neural stimulator.
* Cochlear implant.
* Ocular foreign body (e.g. metal shavings).
* Insulin pump.
* Metal shrapnel or bullet.

When subjects can provide evidence that their implanted device is labeled compatible with MRI, exceptions to the above exclusions can be made and recorded in the note.

Furthermore, certain subject groups will be excluded because of the administration of MRI contrast agents. The weight limit is related to availability of investigational contrast agents. Because of recent concerns about Nephrogenic Systemic Fibrosis/Nephrogenic Fibrosing Dermopathy after gadobenate exposure in patients with end-stage renal disease, renal excretory function will be determined and patients with severe renal excretory dysfunction are excluded from this research protocol.

* Pregnant women (subjects who are uncertain as to whether they are pregnant will be required to have a quantitative serum pregnancy test within 72 hours) or lactating women.
* Subjects who have experienced an allergic reaction to gadolinium-based contrast agents.
* Subjects with hemoglobinopathies.
* Weight greater than 120 kg.
* Subjects with renal disease (eGFR less than 30 ml/min/1.73m(2), or receiving renal replacement therapy).

The creatinine clearance will be estimated in all subjects as an estimated glomerular filtration rate (eGFR) using the abbreviated MDRD Formula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2007-04-05; Primary Completion 2008-11-25 (Actual)

PRIMARY OUTCOMES:
Conspicuity of occluded arteries after contrast exposure.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Farooki A, Narra V, Brown J. Gadofosveset (EPIX/Schering). Curr Opin Investig Drugs. 2004 Sep;5(9):967-76. PMID 15503653
- [Background] Goyen M, Edelman M, Perreault P, O'Riordan E, Bertoni H, Taylor J, Siragusa D, Sharafuddin M, Mohler ER 3rd, Breger R, Yucel EK, Shamsi K, Weisskoff RM. MR angiography of aortoiliac occlusive disease: a phase III study of the safety and effectiveness of the blood-pool contrast agent MS-325. Radiology. 2005 Sep;236(3):825-33. doi: 10.1148/radiol.2363040577. Epub 2005 Jul 14. PMID 16020554
- [Background] Bluemke DA, Stillman AE, Bis KG, Grist TM, Baum RA, D'Agostino R, Malden ES, Pierro JA, Yucel EK. Carotid MR angiography: phase II study of safety and efficacy for MS-325. Radiology. 2001 Apr;219(1):114-22. doi: 10.1148/radiology.219.1.r01ap42114. PMID 11274545